CLINICAL TRIAL: NCT00974272
Title: Effects of Exenatide on Postprandial Hyperlipidemia and Inflammation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Carl T. Hayden VA Medical Center (U.S. Federal Agency)
Responsible Party: Peter D Reaven, MD, Carl T. Hayden VA Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-015
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Type 2 Diabetes Mellitus; Impaired Glucose Tolerance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance | interventions — Exenatide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Experimental)
  Interventions: Drug: Exenatide
- Placebo (Placebo Comparator)
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Exenatide — Single subcutaneous injection (10 μg)
  Other Names: Byetta
  Arms: Exenatide
Other: Normal Saline — Single subcutaneous injection
  Arms: Placebo

SUMMARY:
The primary goal of this study is to determine the acute effects of exenatide on postprandial hypertriglyceridemia. Secondary goals are to determine whether there are additional improvements in postprandial lipids and lipoproteins and whether (by the reduction of hyperglycemia alone or in combination with declines in hyperlipidemia) exenatide reduces the pro-inflammatory potential of the postprandial period.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed type 2 diabetes (within 3 years) on diet or IGT
* Fasting triglyceride levels >140 and < 400 mg/dl and values varying less than 35% between two screening measurements
* Normal liver function tests and white blood cell count

Exclusion Criteria:

* Type 2 Diabetes for > 3 years or HbA1c ≥ 7.5
* Known or suspected Type 1 Diabetes
* Any diabetes medications in the past 3 weeks, TZD in the prior 3 months or prior regular use of insulin
* Creatinine > 2.0 mg/dl or other evidence of active kidney disease
* Hepatic enzyme elevation > 2x normal
* Known Nonalcoholic Fatty Liver Disease
* Malabsorption of fat or other nutrients, severe lactose intolerance or other significant gastrointestinal or pancreatic problems
* Recent history of nausea or vomiting
* Acute bacterial or viral illness or evidence of other active infection in the past 4 weeks
* A prior cardiovascular event, stable or unstable angina or other major illness in the past 6 months
* Current regular use of anti-inflammatory medications or antioxidants, including over the counter medications and high dose salicylates (>1 g/day)
* Any lipid lowering therapy in the prior 3 weeks other than a statin medication. Subjects receiving a statin medication must be on a stable dose for at least 2 months prior to participation.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Triglyceride concentration in serum | Before and up to 8-hours post-injection

SECONDARY OUTCOMES:
serum or plasma lipoproteins, apolipoproteins and inflammatory markers; endothelial function | Before and up to 8 hours post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Reaven, MD, Principal Investigator — Phoenix VA Healthcare System
Locations (1):
- Phoenix VA Medical Center, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Schwartz EA, Koska J, Mullin MP, Syoufi I, Schwenke DC, Reaven PD. Exenatide suppresses postprandial elevations in lipids and lipoproteins in individuals with impaired glucose tolerance and recent onset type 2 diabetes mellitus. Atherosclerosis. 2010 Sep;212(1):217-22. doi: 10.1016/j.atherosclerosis.2010.05.028. Epub 2010 May 25. PMID 20557887
- [Derived] Koska J, Schwartz EA, Mullin MP, Schwenke DC, Reaven PD. Improvement of postprandial endothelial function after a single dose of exenatide in individuals with impaired glucose tolerance and recent-onset type 2 diabetes. Diabetes Care. 2010 May;33(5):1028-30. doi: 10.2337/dc09-1961. Epub 2010 Mar 3. PMID 20200309